CLINICAL TRIAL: NCT05837741
Title: Standard Hypercaloric, Hyperproteic vs Leucine-enriched Oral Supplements in Patients With Cancer-induced Sarcopenia
Brief Title: Leucine-enriched Formulas in Patients With Tumor-induced Sarcopenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Responsible Party: Principal Investigator, Aura Herrera, Principal Investigator, Maimónides Biomedical Research Institute of Córdoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Sarcopenia-Leucina1
Record Dates: First submitted 2023-04-01; First posted 2023-05-01 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Sarcopenia; Cancer
Keywords: Sarcopenia; Cancer
MeSH Terms: conditions — Sarcopenia; Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard hypercaloric, hyperproteic oral supplement (Active Comparator): Patients will receive 2 supplements per day (Standard hypercaloric, hyperproteic oral supplement)
  Interventions: Dietary Supplement: Standard hypercaloric hyperproteic oral nutritional supplement
- Leucin-enriched hypercaloric, hyperproteic oral supplement (Active Comparator): Patients will receive 2 supplements per day (Leucin-enriched hypercaloric, hyperproteic oral supplement)
  Interventions: Dietary Supplement: Leucine-enriched hypercaloric hyperproteic oral nutritional supplement

INTERVENTIONS:
Dietary Supplement: Standard hypercaloric hyperproteic oral nutritional supplement — Patients will receive nutritional support with Standard hypercaloric hyperproteic oral nutritional supplement
  Arms: Standard hypercaloric, hyperproteic oral supplement
Dietary Supplement: Leucine-enriched hypercaloric hyperproteic oral nutritional supplement — Patients will receive nutritional support with Leucine-enriched hypercaloric hyperproteic oral nutritional supplement
  Arms: Leucin-enriched hypercaloric, hyperproteic oral supplement

SUMMARY:
Currently there is a lack of evidence for recommending specific oral supplements (OS) for nutritional support in patients with cancer, including leucine-enriched supplements.

DETAILED DESCRIPTION:
Appropriate clinical trials that compare anthropometric and biochemical changes in nutritional parameters and clinical outcomes in patients with cancer-induced sarcopenia are required

ELIGIBILITY:
Inclusion Criteria:

* patients of both sexes, age > 18 y-old
* cancer of different origin treated with systemic treatment chemo, radiotherapy or combination treatment t
* weight loss >5% during the previous three months or >10% during the previous six months

Exclusion Criteria:

* end-stage kidney disease
* life expectancy < 2 weeks

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Muscle mass gain | 3 Months
  Changes in Muscle mass (%) determined by BIA and echography

SECONDARY OUTCOMES:
Fat mass change | 3 Months
  Changes in fast mass (%) determined by BIA and echography
Phase angle change | 3 Months
  Changes in phase angle determined by BIA
Changes in albumin | 3 Months
  Changes in serum albumin levels (g/dL)
Changes in prealbumin | 3 Months
  Changes in serum prealbumin levels (mg/dL)
Changes in CRP | 3 Months
  Changes in serum CRP levels (g/L)

CONTACTS AND LOCATIONS:
Overall Officials: Aura D Herrera Martinez, PhD, Principal Investigator — IMIBIC-HURS
Locations (1):
- IMIBIC, Córdoba, Cordoba, Spain

IPD SHARING:
Plan to Share IPD: No